CLINICAL TRIAL: NCT05375812
Title: NIH Investigative Deep Phenotyping Study of Gulf War Veteran Health (Project NIH IN-DEPTH)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000051; 000051-N
Record Dates: First submitted 2022-05-13; First posted 2022-05-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-18

CONDITIONS: Gulf War Illness
Keywords: Veteran; Gwi (Gulf War Illness); Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GWI: Gulf War Veterans
- HVC: Healthy Volunteer Controls

SUMMARY:
Background:

Gulf War illness (GWI) affects up to 210,000 U.S. veterans who served in the Middle East during the Gulf War in 1990-1991. Symptoms include fatigue, muscle and joint pain, forgetfulness, headaches, rashes, and sleep disturbances. Routine exams cannot determine the cause of GWI. Researchers need more information to understand this disease.

Objective:

This natural history study will look for differences in Gulf War veterans who experienced GWI and those who did not.

Eligibility:

Gulf War veterans with GWI. Healthy Gulf War veterans who do not have GWI are also needed.

Design:

Participants will stay in the NIH Clinical Center as an inpatient for 2 weeks. They will undergo many tests.

Blood will be drawn many times throughout the study. Participants will also give urine, saliva, and stool samples.

Scans to measure the brain, leg muscles, bone density and body mass will be done.

They will have an exercise stress test and muscle strength tests.

They will have a sleep study. They will have tests to look at how well the brain, heart and lungs are working.

Participants will sleep in a specialized room that measures the amount of oxygen they use and the carbon dioxide they produce on four consecutive nights.

A sample of fluid will be collected from inside the spine.

Participants will take many surveys. Some will ask about their activities. Some will be about emotional and mental health. Some will be about thinking, memory, and behavior.

Optional tests include other imaging scans and testing the autonomic nervous system. Samples of skin and muscle may be taken.

After discharge, participants will wear activity monitors for 14 days. They will keep a diary of their symptoms, including fatigue, pain, and sleep, while wearing the monitors.

DETAILED DESCRIPTION:
Study Description:

This protocol is part of a joint collaboration with the Veterans' Administration (VA) known as (Project IN-DEPTH). The Veterans' Administration protocol will recruit and identify participants for the NIH study, and maintain a repository of data and samples through a VA protocol (VA IN-DEPTH). The NIH protocol (NIH IN-DEPTH) will conduct deep phenotyping evaluations on study participants.

Gulf War Illness (GWI) and Gulf War Chronic Multi-Symptom Illness are names that have been used to describe a disorder of fatigue, muscle and joint pain, loss of concentration, forgetfulness, headache, respiratory complaints, rashes, sleep disturbances, and/or gastrointestinal distress. The purpose of this study is to learn more about GWI from veterans deployed in Persian Gulf during the first Gulf War.

In this study, two groups of veterans who were deployed to the Persian Gulf war between August 1990 and June 1991 will be enrolled: those who are healthy veteran controls (HVC) and those with GWI. Participants will have an inpatient study visit typically lasting 14 days to explore clinical and biological phenotypes through evaluations via questionnaires, medical procedures such as exercise testing, history and physical examination, and laboratory evaluation of samples.

This protocol is a "sister study" to the NIH protocol 16-N-0058: Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) at NIH. The symptoms of GWI and ME/CFS are very similar and much may be learned about each disorder through comparison. For this reason, the two studies will use similar methods. Participants in 16-N-0058 had previously consented to sharing of data, therefore datasets from this NIH IN-DEPTH protocol and 16-N-0058 will be shared and combined to perform several of the planned exploratory analyses.

This study will take place at the National Institutes of Health (NIH) Clinical Center in Bethesda, Maryland.

Objectives: Primary Objective:

To explore and compare the clinical and biological phenotypes of veterans with GWI and healthy veteran controls (HVC) at baseline.

Exploratory Objectives:

To explore the pathophysiology of fatigue and GWI symptom flares. Fatigue will be explored using tasks designed to create muscular and cognitive fatigue. GWI symptom flares will be explored using an exercise stress test and measuring the symptomatic and biological changes.

To compare the clinical and biological phenotypes between GWI, HVC, ME/CFS, and healthy volunteers.

Endpoints: Outcome measures

The primary purpose of this protocol is to perform exploratory analysis of collected data and samples for the generation of new hypotheses regarding GWI. The types of analyses to be performed will be wide ranging. Planned areas of focus may include:

* Characterization of the immune system and inflammatory signaling.
* Characterization of the pattern of microbiome.
* Characterization of bioenergetics, autonomic, and metabolic function.
* Characterization of neurocognition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for all veterans:

* Ability to provide informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 48-70 at time of enrollment into VA IN-DEPTH Study
* Veterans who were deployed to Gulf Region ODS/S between August 1990 - June 1991.
* Self-reported completion of at least the seventh grade of school.
* Fluency in speaking, reading, and understanding English.
* Underwent screening as part of the VA IN-DEPTH study and were unanimously determined to be eligible by the IN-DEPTH Adjudication Committee.
* Agree not to smoke in the 4 hours prior to CPET procedure

EXCLUSION CRITERIA:

Exclusion criteria for all veterans:

* Current or past psychotic disorder including depression with psychosis, bipolar disorder with psychotic symptoms and schizophrenia
* Current DSM-5-defined major depression disorder, generalized anxiety disorder, posttraumatic stress disorder, panic disorder, or obsessive-compulsive disorder unless managed for more than six months with a stable treatment regimen
* Current or past substance use disorder within last five years as diagnosed on the Structured Clinical Interview for DSM-5 (SCID-5). Prior or prescription marijuana use within the past five years will not be an exclusion.
* Current suicidal ideation
* History of head injury leading to moderate or severe traumatic brain injury, as detailed by loss of consciousness for greater than 30 minutes, a Glasgow Coma Score of 12 or less at the time of injury, post-traumatic amnesia greater than one day, or brain-scan changes related to a head injury. Persons having a history of mild TBI (mTBI) will not be excluded.
* Women who are pregnant, breastfeeding, or are within one-year post-partum.
* Current or previous malignancy. A history of malignancy that has fully resolved with surgical resection only (e.g. no chemotherapy, radiation therapy, or immunotherapy) will be allowed.
* Current systemic immunologic disorders (e.g. Type 1 diabetes, rheumatoid arthritis). Local immunological disorder (e.g. atopic dermatitis, stable autoimmune thyroid disease) and allergic disorders will be allowed.
* Current or previous long-term immune suppressive therapy. Systemic steroid use, even short-term, must not have been used within the month prior to enrollment
* Any medical condition that would make the study procedures risky for the participant (e.g. congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, severe osteoarthritis, exercise-induced angina and poorly controlled asthma).
* Active participation in a clinical protocol (e.g. anti-inflammatory drug intervention study) which includes an intervention that may affect the results of the current study.
* Inability to perform the bicycling exercise task. (e.g. coronary artery disease, not having a lower limb, disabling stroke)
* Not willing to allow for research data and samples to be shared broadly with other researchers.
* Symptom severity that makes it impossible for the volunteer to travel to NIH for extended inpatient evaluation
* Use of medications with a high-risk for withdrawal-related complications (i.e. long-acting opiates or benzodiazepines).

Additional Exclusion criteria for participants undergoing TMS:

- Pacemaker, implanted pump, stimulator, cochlear implant or metal objects inside the eye or skull.

Participants with unconfirmed metal may have further evaluation to rule out metal in the eye or skull.

Participants without metal after evaluation may proceed to TMS.

- A personal history of seizure disorder

Additional Exclusion criteria for participants undergoing MRI:

- Metal in the body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or having a history of being a welder or metal worker, since small metal fragments may be in the eye. Participants with unconfirmed metal may have further evaluation to rule out metal in the eye

or skull. Participants without metal after evaluation may proceed to MRI.

* Substantial claustrophobia
* Inability to lie on back for up to 2 hours

Additional Exclusion criteria for Healthy Veteran Controls:

- Meets modified Kansas criteria for GWI.

Ages: 48 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A Target of 50 GWI participants and 25 Healthy volunteer controls will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To explore and compare the clinical and biological phenotypes of veterans with GWI and healthy veteran controls (HVC) at baseline. | one time visit
  Evaluate a number of clinical and biological measures.

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Walitt, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000051-N.html